CLINICAL TRIAL: NCT01116661
Title: A Phase 2 Study of Aminolevulinic Acid (ALA) to Enhance Visualization and Resection of Tumors of the Brain
Brief Title: Safety Study of Aminolevulinic Acid (ALA) to Enhance Visualization and Resection of Tumors of the Brain
Acronym: ALA
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: The primary objective for high grade gliomas has been met and the FDA has now approved the drug (Gleolan) for use in the United States.
Sponsor: University of California, San Francisco (Other)
Responsible Party: Principal Investigator, Mitchel Berger, MD, Chairman, University of California, San Francisco
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 10101
Record Dates: First submitted 2010-05-03; First posted 2010-05-05 (Estimated); Results first posted 2019-05-29 (Actual); Last update posted 2019-05-29 (Actual); Status verified 2019-05

CONDITIONS: Glioma
Keywords: glioma; high grade glioma, low grade glioma
MeSH Terms: conditions — Glioma

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- ALA for glioma (WHO G1-IV) subjects (Experimental): Up to 300 patients with diagnosed glioma (WHO G1-IV) eligible for surgery will be entered into the trial and will be given 5-Aminolevulinic Acid (ALA) orally at a dose of 20mg/kg body weight preoperatively
  Interventions: Drug: 5-Aminolevuline Acid (ALA)

INTERVENTIONS:
Drug: 5-Aminolevuline Acid (ALA) — Given orally at a dose of 20 mg/kg body weight 3hrs before anesthesia prior to surgery

SUMMARY:
The prodrug, 5-Aminolevulinic acid (ALA), has been shown to lead to intracellular accumulation of fluorescent porphyrins in high grade malignant gliomas in the brain. On imaging, this accumulation of fluorescent porphyrins helps delineate tumor borders, resulting in the surgeon being better able to visualize and thus able to make a complete, or near-complete resection of the tumor.

DETAILED DESCRIPTION:
The drug, 5-aminolevulinic acid (ALA), which leads to intracellular accumulation of fluorescent porphyrins in gliomas will be used under investigation for identification and resection of high and low grade gliomas. Surgery will be done using a modified neurosurgical microscope, with a fluorescent kit that enables switching from the conventional white light to a violet-blue excitation light for visualization during tumor resection. If deemed safe by the neurosurgeon, any area of the resection bed determined to be fluorescence-positive for tumor will be removed with appropriate designation of tissue for histopathological evaluation. After this resection, additional fluorescence images will be obtained and the process repeated until the image is negative for tumor. At all times, the decision to resect will be limited by clinical judgment of safety.

The desire is that a more complete resection will occur due to the surgeon's ability to better visualize and distinguish between tumor and normal tissue, and thus be able to remove as much, or most of, the tumorous tissue, resulting in a better outcome for the patient, or for future patients.

ELIGIBILITY:
Inclusion Criteria:

1. Presumptive diagnosis of high grade or low grade glioma based on imaging studies, or will have recurrent high-grade or low grade gliomas that have previously undergone diagnosis (astrocytoma, oligodendroglioma, mixed oligo-astrocytoma, anaplastic astrocytoma, and glioblastoma multiforme). Both of these groups will be undergoing craniotomy for tumor resection.
2. Patient age 18 to 72 years.
3. Karnofsky performance of 60% or greater
4. Patients must have normal organ and marrow function as defined below:

   Leukocytes >3,000/μL Absolute neutrophil count >1,500/μL Platelets >100,000/μL Total bilirubin within normal institutional limits AST (SGOT)/ALT (SGPT) <2.5 X institutional upper limit of normal Creatinine within normal institutional limits or Creatinine clearance ≥60 mL/min/1.73 m2 for patients with creatinine levels above institutional normal.
5. The effects of Aminolevulinic Acid (ALA) on the developing human fetus are unknown. Therefore, women of child-bearing potential and men must agree to use adequate contraception (hormonal or barrier method of birth control; abstinence) prior to study entry and for the duration of study participation.
6. Patient must have the ability to understand and the willingness to sign a written informed consent document or have a parent or guardian with the ability to understand and the willingness to sign the written informed consent.

Exclusion Criteria:

1. Subjects with a history of allergic reactions attributed to compounds of similar chemical or biologic composition to aminolevulinic acid (ALA).
2. Subjects with a history or family history of Porphyrias
3. Subjects with uncontrolled intercurrent illness including, but not limited to ongoing or active infection, symptomatic congestive heart failure, unstable angina pectoris, cardiac arrhythmia, or psychiatric illness/social situations that would limit compliance with study requirements.
4. Pregnancy.

Ages: 18 Years to 72 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 199 (Actual)
Dates: Start 2010-08 (Actual); Primary Completion 2017-12-28 (Actual); Study Completion 2019-02-28 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Mitchel S Berger, MD, Principal Investigator — UCSF Department of Neurosurgery
Locations (1):
- UCSF Department of Neurosurgery, San Francisco, California, United States

REFERENCES:
- [Derived] Widhalm G, Olson J, Weller J, Bravo J, Han SJ, Phillips J, Hervey-Jumper SL, Chang SM, Roberts DW, Berger MS. The value of visible 5-ALA fluorescence and quantitative protoporphyrin IX analysis for improved surgery of suspected low-grade gliomas. J Neurosurg. 2019 May 10;133(1):79-88. doi: 10.3171/2019.1.JNS182614. Print 2020 Jul 1. PMID 31075771

RESULTS

PARTICIPANT FLOW:
Groups:
- Single Dose ALA for Newly Diagnosed and Recurrent HGG: 5-Aminolevuline Acid: Given orally at a dose of 20 mg/kg body weight 3hrs before anesthesia prior to surgery for both newly diagnosed and recurrent High grade gliomas
Period: Overall Study
Arm/Group | Single Dose ALA for Newly Diagnosed and Recurrent HGG
Started | 199
Completed | 197
Not Completed | 2

BASELINE CHARACTERISTICS:
Population: The analysis population is the same as the assignment in Participant flow
Groups:
- 5 - Aminolevuline Acid in Patients With HGG: 5-Aminolevuline Acid: Given orally at a dose of 20 mg/kg body weight 3hrs before anesthesia prior to surgery
Arm/Group | 5 - Aminolevuline Acid in Patients With HGG
Number analyzed (Participants) | 197
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | NA — Study did not allow for participates under 18 years of age
  Between 18 and 65 years | 160
  >=65 years | 37
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 78
  Male | 119
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 9
  Native Hawaiian or Other Pacific Islander | 2
  Black or African American | 0
  White | 162
  More than one race | 0
  Unknown or Not Reported | 24
Region of Enrollment [Number; unit: participants]
  United States | 197

OUTCOME MEASURES:

1. Primary Outcome: The Percentage of Biopsies Taken From the Most Fluorescent Tissues That Have Tumorous Content.
Description: Biopsies were examined by a pathologist to determine the amount of tumor content from the most fluorescent tissues
Time Frame: 1 day
Population: All patient who received 5-Aminolevuline Acid prior to surgical resection
Measure: Median (95% Confidence Interval); unit: percentage of biopsies
Groups:
- 5- Aminolevuline Acid Given to HGG Participants: 5-Aminolevuline Acid: Given orally at a dose of 20 mg/kg body weight 3hrs before anesthesia prior to surgery
Arm/Group | 5- Aminolevuline Acid Given to HGG Participants
Number analyzed (Participants) | 197
percentage of biopsies | 90.9 [9.9 to 100]

2. Secondary Outcome: Number of Participants With Adverse Events
Description: Number of Participants with Adverse Events, as defined by grade 3 to 5 AEs and SAEs related to study drug. .
Time Frame: 14 days
Population: Patients who received study drug
Measure: Count of Participants; unit: Participants
Arm/Group | 5- Aminolevuline Acid Given to HGG Participants
Number analyzed (Participants) | 197
Participants | 14

ADVERSE EVENTS:
Time Frame: From time of ALA dosing up to 14 days post- operative
Arm/Group | 5- Aminolevuline Acid Given to HGG Participants
All-Cause Mortality (participants affected / at risk) | 59/199
Serious Adverse Events (participants affected / at risk) | 12/199
Other Adverse Events (participants affected / at risk) | 25/199
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | 5- Aminolevuline Acid Given to HGG Participants (N=199)
Hypotension (Cardiac disorders) | 1 (1)
Intracranial hemorrhage (Nervous system disorders) | 1 (1)
Infection - with Grade 3 or 4 nuetrophils (Infections and infestations) | 1 (2)
Infection - other (Infections and infestations) | 1 (1)
Hyponatremia (Metabolism and nutrition disorders) | 2 (2)
Mental status (Nervous system disorders) | 1 (1)
Seizure (Nervous system disorders) | 4 (4)
thrombosis/embolism (Vascular disorders) | 1 (1)
Vascular - other (Vascular disorders) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | 5- Aminolevuline Acid Given to HGG Participants (N=199)
Lymphopenia (Blood and lymphatic system disorders) | 3 (4)
Photosensitivity (Skin and subcutaneous tissue disorders) | 5 (8)
Dermatology/skin (Skin and subcutaneous tissue disorders) | 3 (3)
Dry Skin (Skin and subcutaneous tissue disorders) | 1 (1)
Flushing (Skin and subcutaneous tissue disorders) | 1 (1)
ALT,SGPT increase (Metabolism and nutrition disorders) | 2 (2)
Alkaline Phosphatase (Metabolism and nutrition disorders) | 1 (1)
AST,SGOT increase (Metabolism and nutrition disorders) | 1 (1)
Hyperbilirubinemia (Metabolism and nutrition disorders) | 1 (1)
Hemoglobin decrease (Blood and lymphatic system disorders) | 1 (1)
Hypotension (Cardiac disorders) | 2 (2)
hypertension (Cardiac disorders) | 1 (1)
Fatigue (General disorders) | 1 (1)
Pain - skin (Skin and subcutaneous tissue disorders) | 1 (1)
metabolic/Laboratory - other (Metabolism and nutrition disorders) | 3 (3)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2013-03-14): https://cdn.clinicaltrials.gov/large-docs/61/NCT01116661/Prot_SAP_000.pdf